CLINICAL TRIAL: NCT07129577
Title: Point of Care Testing in Emergency Departments After Mild Traumatic Brain Injury (POCkET)
Brief Title: Point of Care Testing in Emergency Departments After Mild Traumatic Brain Injury
Acronym: POCkET
Status: Not yet recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Virginia Newcombe, Honorary Consultant in Critical Care and Emergency Medicine / Clinician Scientist Fellow, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: IRAS 353032
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Injuries, Head; Traumatic Brain Injuries
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Traumatic brain injury (TBI) is estimated to have the highest incidence of all common neurological disorders, affecting 50 to 60 million people worldwide each year. In the UK, approximately one million people attend an Emergency Department (ED) annually following a head injury, and 80-90% of these are classified as mild TBI (mTBI), also referred to as concussion. In the acute setting, mTBI is typically defined by a Glasgow Coma Scale (GCS) score of 13-15 on presentation.

Current acute management focuses primarily on identifying which patients require a CT head scan to detect life threatening injuries that may need neurosurgical intervention, observation, or neurocritical care. However, there is increasing recognition that the term "mild" can be misleading. Many patients, including those with normal CT scans,experience persistent functional, cognitive, and symptomatic deficits that may benefit from further intervention and follow-up care.

Blood biomarkers offer significant potential to improve the early diagnosis, risk stratification, and prognostication of mTBI in the ED setting. While these biomarkers are increasingly being developed and evaluated in moderate and severe TBI, their clinical utility in mild TBI has not yet been definitively demonstrated.

To fully assess their potential value, it is essential to understand the current care pathways for mTBI in the ED, how they are implemented in practice, and where biomarker information could meaningfully enhance clinical decision making and improve patient outcomes.

The POCKET study will use a systems engineering approach, in combination with health economic evaluation, to assess the potential role and utility of point-of-care blood biomarkers in the management of mild TBI in UK emergency departments. This research will be conducted using the Abbott biomarker platform.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age)
* Glasgow Coma Score >12
* Presentation within 24 hours of head injury
* Meet criteria to be assessed using NICE NG232 clinical decision support tool (CDST).
* Patients with a prior history of TBI may still be included.

Exclusion Criteria:

* Participant without capacity and no available patient legal representative or professional consultee.
* Participant with capacity unwilling to provide informed consent
* Unable to adequately understand written and verbal English.
* Prisoners currently in custody of HM Prison Service

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to Emergency Departments (EDs) with mild traumatic brain injury (mTBI) defined as Glasgow Coma Score >12.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Understanding of the current clinical pathway and how use of point of care biomarkers may change this. | From enrolment to 6 months

IPD SHARING:
Plan to Share IPD: Undecided